CLINICAL TRIAL: NCT06933654
Title: Iris Suture Fixation vs Iris Claw for Aphakic Correction
Brief Title: Iris Suture Fixation vs Iris Claw for Correction of Aphakia
Acronym: IOLs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Benha University (Other)
Collaborators: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Ehab Mohamed Elsayed Mohamed Saad, Lecturer, Benha University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: aphakic correction; Benha University (Other: Al-Azhar University)
Record Dates: First submitted 2025-04-11; First posted 2025-04-18 (Actual); Last update posted 2025-04-18 (Actual); Status verified 2025-04

CONDITIONS: Aphakic Eye
Keywords: Iris suture fixation , iris claw, aphakia
MeSH Terms: conditions — Aphakia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Iris claw IOL) (Active Comparator): included 25 eyes in which the iris claw lens was used, the lens used in this study was the Artisan aphakia IOL (Ophtec BV, Groningen, The Netherlands) which is a PMMA IOL with an 8.5 mm length, 1.04-mm maximum height and 5.4-mm optical zone width.
  Interventions: Procedure: IOL implantation surgery for aphkic eye
- Group B (Iris fixation IOL) (Active Comparator): included 25 eyes were subjected to iris fixation of posterior chamber foldable IOLs. eyes in which a single piece PMMA IOL was implanted. The IOL is 6 mm optic, 12.75 mm overall diameter, and has one eyelet for suture fixation in each haptic. A constant was 118.2.
  Interventions: Procedure: IOL implantation surgery for aphkic eye

INTERVENTIONS:
Procedure: IOL implantation surgery for aphkic eye — Aphakic eyes underwent secondary intraocular lens (IOL) implantation using one of two techniques. In Group A, an iris-claw IOL (Artisan aphakia IOL, Ophtec BV, The Netherlands) was implanted and fixated to the mid-peripheral iris via enclavation. In Group B, a posterior chamber foldable PMMA IOL was fixated to the iris using transscleral sutures passed through eyelets in the haptics. All procedures were performed under peribulbar anesthesia using standard aseptic technique, and postoperative management included topical antibiotics and corticosteroids.

SUMMARY:
Evaluate and compare the advantages and disadvantages of iris suture fixation versus iris claw of posterior chamber IOLs

DETAILED DESCRIPTION:
The eyes were randomly divided into two groups, A and B. Group A included 25 eyes in which an iris claw lens was used; specifically, the Artisan aphakia intraocular lens (Ophtec BV, Groningen, The Netherlands), a PMMA IOL with an 8.5 mm length, 1.04 mm maximum height, and a 5.4 mm optical zone width. Group B also included 25 eyes, in which iris fixation of posterior chamber foldable IOLs was performed using a single-piece PMMA IOL. This IOL had a 6 mm optic, a total diameter of 12.75 mm, and featured one eyelet for suture fixation in each haptic. The A-constant used was 118.2.

ELIGIBILITY:
Inclusion Criteria:

* Surgical aphakia with no capsular support, with CDVA 4/60 or better on Snellen chart including: Aphakic eyes after complicated cataract surgery, crystalline lens subluxation (Marfan syndrome, pseudoexofoliation syndrome or trauma), 2nd intervention in traumatized eyes, cases with sublaxated or dislocated IOLs.

Exclusion Criteria:

* Surgical aphakia with decompensated corneas, aphakic patients with posterior segment pathologies like cystoid macular edema, choroidal neovascular membrane, aphakic patients with insufficient iris tissue, and rubeosis iridis, aphakic patients with intractable glaucoma.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2024-04-01 (Actual); Primary Completion 2024-11-30 (Actual); Study Completion 2024-12-01 (Actual)

PRIMARY OUTCOMES:
Best-corrected visual acuity (BCVA) | at 6 months postoperatively
  BCVA in logMAR , to evaluate and compare visual recovery between the iris-claw and iris suture-fixated IOL groups.

CONTACTS AND LOCATIONS:
Overall Officials: Ehab Saad, Lecturer, Principal Investigator — Benha University, Ebsar Eye Center
Locations (1):
- Ebsar Eye Center, Cairo, Egypt